CLINICAL TRIAL: NCT00355836
Title: Can Motor Imagery Enhance Recovery of Hand Function After Stroke? Evaluation of Motor Imagery Training.
Brief Title: Recovery of Hand Function Through Mental Practice.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CZH/4/153
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Stroke
Keywords: Motor Imagery; Stroke; Neuro-rehabilitation; health psychology; neuroscience; randomised controlled trial
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Behavioral: Mental Imagery

SUMMARY:
The purpose of this study is to assess the therapeutic benefits of motor imagery training in stroke patients with persistent motor weakness.

DETAILED DESCRIPTION:
Stroke is a common and highly debilitating illness. Many patients (41-45%) experience chronic motor impairments (Dijkerman et al., 1996) and limitations in activities of daily living (Wade & Langton Hewer, 1987) even after extensive neurological rehabilitation. They often result in long-term dependence at a considerable cost to the carers and the health service. It is therefore crucial to optimise motor recovery after stroke. This study investigates the therapeutic benefits of motor imagery training in stroke patients with a motor weakness.

Evidence for the idea that motor imagery training could enhance the recovery of hand function comes from several separate bases of evidence: the sports literature; neurophysiological evidence; evidence from health psychology research; as well as preliminary findings using motor imagery techniques in stroke patients.

There is evidence to suggest that mental rehearsal of movement can produce effects normally attributed to practising the actual movements. Imagining hand movements could stimulate the redistribution of brain activity, which accompanies recovery of hand function, thus resulting in a reduced motor deficit. Patients are assessed before and after a four-week evaluation period. In this randomised controlled trial 45 patients daily mentally rehearse movements with their affected hand under close supervision. Their recovery is compared to 45 patients who perform closely supervised non-motor mental rehearsal, and 45 patients who are not engaged in a training program.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of stroke in the last 1-6 months Persisting upper limb weakness -

Exclusion Criteria:

Alcohol/ Drug abuse Psychiatric history Previous illness that has impacted on individuals Activity of Daily living

- Dementia (assessed by MSQ) Severe Aphasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) (Lyle, 1981)

SECONDARY OUTCOMES:
Grip strength (dynamometer; Heller et al., 1987),
Nine hole pegboard task (Mathiowetz et al., 1985, Wade [ref]),
Function Limitation Profile
Barthel Index
Recovery Locus of Control

CONTACTS AND LOCATIONS:
Overall Officials: Marie Johnston, Prof, Principal Investigator — University of Aberdeen
Locations (2):
- United Kingdom (2):
  - University of Aberdeen, Aberdeen
  - Ninewells Hospital, Dundee